CLINICAL TRIAL: NCT06079411
Title: Low-Cost Virtual Therapeutics and Digital Biomarkers for the Early Assessment and Personalized Treatment of Mild Cognitive Impairment
Brief Title: Virtual Therapeutics for MCI
Acronym: VR-MCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Istituto Superiore di Sanità (Other); University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 39M202
Record Dates: First submitted 2023-09-26; First posted 2023-10-12 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAU (Active Comparator): the treatment as usual (TAU; i.e., visuospatial "paper and pencil" stimulation) will consist of "paper and pencil" exercises used in clinical routine of 8 sessions of 30/40 minutes 3 times a week.
  Interventions: Other: treatment as usual
- VR non-embodied (Experimental): the non-embodied spatial training will consist of egocentric and allocentric spatial memory training with passive navigation of 8 sessions of 30/40 minutes 3 times a week.
  Interventions: Device: virtual reality non-embodied
- VR embodied (Experimental): the embodied spatial training will consist of egocentric and allocentric spatial memory training with active navigation of 8 sessions of 30/40 minutes 3 times a week.
  Interventions: Device: virtual reality embodied

INTERVENTIONS:
Device: virtual reality non-embodied — the non-embodied virtual reality spatial training will consist of egocentric and allocentric spatial memory training with passive navigation of 8 sessions of 30/40 minutes 3 times a week.
  Arms: VR non-embodied
Device: virtual reality embodied — the embodied virtual reality spatial training will consist of egocentric and allocentric spatial memory training with active navigation of 8 sessions of 30/40 minutes 3 times a week.
  Arms: VR embodied
Other: treatment as usual — the treatment as usual (TAU; i.e., visuospatial "paper and pencil" stimulation) will consist of "paper and pencil" exercises
  Arms: TAU

SUMMARY:
Mild Cognitive Impairment (MCI) is a term used to describe the transitional stage that occurs between normal aging and the onset of dementia. Spatial disorientation is often considered a significant indicator for diagnosing dementia. Numerous studies have documented deficits in both the allocentric and egocentric spatial frames of reference, as well as difficulties in transitioning between them, in individuals with MCI. Rapid advances in computing technology have enabled researchers to conduct cognitive training and rehabilitation interventions with the assistance of technology. Therefore, the aim of the study is to use virtual therapeutics to train MCI spatial memory.

DETAILED DESCRIPTION:
The current study aims to design, develop and test virtual therapeutics to train MCI spatial memory through virtual reality rehabilitation. 36 Participants will be randomly assigned to three different conditions: embodied low-end spatial VR training vs. the treatment as usual (TAU; i.e., visuospatial "paper and pencil" stimulation) vs. a non-embodied low-end spatial VR training. The three conditions will consist of at least 8 sessions of 30/40 minutes 3 times a week.

The study will measure changes in spatial memory, in particular in egocentric and allocentric memory. Each patient will be tested 3 times: 3 weeks before the pre-test (control waiting period), at the pre-test and after the intervention, namely post-test (3 time points).

ELIGIBILITY:
Inclusion Criteria:

* a change in cognition recognized by patients or observers (Caregiver/examiner)
* an objective impairment in one or more cognitive domains using traditional neuropsychological tests;
* autonomy or slight dependence on daily life activities;
* absence of diagnosis of dementia
* absence of cognitive impairment measured by the mini-mental state examination;
* aged 65 or over

Exclusion Criteria:

* the presence of acute stroke/transient ischemic attack occurred in the 6 months prior to the enrollment visit;
* the presence of aphasia and/or neglect;
* the presence of other concomitants severe neurological/psychiatric diseases (e.g., hemiparesis, multiple system atrophy, muscular skeletal/orthopedic deficits that limit movement)
* the presence of physical and/or functional deficits;
* the comorbidity with severe neurological and/or psychiatric diseases (e.g., neoplasms, multiple sclerosis, amyotrophic lateral sclerosis, Huntington's disease, schizophrenia, addiction, personality disorder, eating disorder) or with psychiatric conditions not under drug treatment (anxiety-depressive syndrome, bipolarism);
* the history of head trauma with loss of consciousness
* recurrent vertigo.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The long-term visuospatial memory scores from Corsi supra span | change from waiting list to pre-test (after 3 weeks from waiting list) and post-test (after 6 weeks from waiting list) and change from pre-test to post-test (after 3 weeks from pre-test)
  A lower Corsi supra span score represents a lower visuospatial memory. The minimum score is 0.06 and the maximum is 29.16. Scores will be corrected for age and education and they depend on the score of the Corsi Block Tapping Test.
the spatial rotation score from the Manikin Test | change from waiting list to pre-test (after 3 weeks from waiting list) and post-test (after 6 weeks from waiting list) and change from pre-test to post-test (after 3 weeks from pre-test)
  A lower score in The Manikin test represents lower spatial rotation ability. The minimum score is 0, and the maximum score is equal to 30.

SECONDARY OUTCOMES:
the cognitive global scores from Mini Mental State Examination | change from waiting list to pre-test (after 3 weeks from waiting list) and post-test (after 6 weeks from waiting list) and change from pre-test to post-test (after 3 weeks from pre-test)
  A lower score in Mini Mental State Examination represents a worse symptom severity. The minimum score is 0, and the maximum score is equal to 30. Scores will be corrected for age and education.
The verbal memory scores from the Babcock test | change from waiting list to pre-test (after 3 weeks from waiting list) and post-test (after 6 weeks from waiting list) and change from pre-test to post-test (after 3 weeks from pre-test)
  A lower score in the Babcock test represents a worse symptom severity. The minimum score is 0, and the maximum score is equal to 8 for the immediate score; The minimum score is 0, and the maximum score is equal to 8 for the delayed score. Scores will be corrected for age and education
The short term visuospatial memory scores from the Corsi Block Tapping Test- Forward | change from waiting list to pre-test (after 3 weeks from waiting list) and post-test (after 6 weeks from waiting list) and change from pre-test to post-test (after 3 weeks from pre-test)
  A lower score in the Corsi Block Tapping Test- Forward represents a worse symptom severity. The minimum score is 3, and the maximum score is equal to 9. Scores will be corrected for age and education.
the visuospatial working memory scores from the Corsi Block Tapping Test- Backward | change from waiting list to pre-test (after 3 weeks from waiting list) and post-test (after 6 weeks from waiting list) and change from pre-test to post-test (after 3 weeks from pre-test)
  A lower score in the Corsi Block Tapping Test- Backward represents a worse symptom severity. The minimum score is 3, and the maximum score is equal to 8. Scores will be corrected for age and education.
The attention and executive functions score from the Trail Making Test | change from waiting list to pre-test (after 3 weeks from waiting list) and post-test (after 6 weeks from waiting list) and change from pre-test to post-test (after 3 weeks from pre-test)
  A higher score in the Trail Making Test represents a worse symptom severity. The minimum score is 0 and no time limit for the maximum score for Trail Making Test part A, Trail Making Test part B and Trail Making Test part BA scores.
the visuospatial score from the Clock Drawing Test | change from waiting list to pre-test (after 3 weeks from waiting list) and post-test (after 6 weeks from waiting list) and change from pre-test to post-test (after 3 weeks from pre-test)
  A lower score in the Clock Drawing Test represented a worse symptom severity. The minimum score is 0, and the maximum score is equal to 13.
the spatial rotation score from the Money Roadmap test | change from waiting list to pre-test (after 3 weeks from waiting list) and post-test (after 6 weeks from waiting list) and change from pre-test to post-test (after 3 weeks from pre-test)
  A lower score in the Money Roadmap test represented a worse symptom severity. The minimum score is 0, and the maximum score is equal to 32.
Subjective Subjective Spatial Navigation Complaints sub-scale number 7 | change from waiting list to pre-test (after 3 weeks from waiting list) and post-test (after 6 weeks from waiting list) and change from pre-test to post-test (after 3 weeks from pre-test)
  A higher score in Subjective Spatial Navigation Complaints represented a worse symptom severity. The minimum score is 0, and the maximum score is 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Milan, Lombardy, Italy